CLINICAL TRIAL: NCT01379300
Title: A Randomized Clinical Trial to Validate Novel Biomarker Approaches After Single Doses of Anticoagulants in Healthy Young Male Subjects and in Healthy Elderly Subjects
Brief Title: A Study to Investigate Biomarkers After Single Doses of Anticoagulants in Healthy Young Male and Healthy Elderly Participants (MK-0000-216 AM1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0000-216
Record Dates: First submitted 2011-06-03; First posted 2011-06-23 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Thrombosis
Keywords: Hemophilia B
MeSH Terms: conditions — Thrombosis; Hemophilia B | interventions — Dabigatran; Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dabigatran (Experimental): Single 150-mg dose of dabigatran etexilate
  Interventions: Drug: dabigatran etexilate
- Rivaroxaban (Experimental): Single 20-mg dose of rivaroxaban
  Interventions: Drug: rivaroxaban
- No intervention (No Intervention): No study drug will be administered

INTERVENTIONS:
Drug: dabigatran etexilate — dabigatran etexilate, orally, as 2 x 75-mg capsules (150 mg), single administration
  Arms: Dabigatran
Drug: rivaroxaban — rivaroxaban, orally, as 2 x 10-mg tablets (20 mg), single administration
  Arms: Rivaroxaban

SUMMARY:
This is a study to investigate biomarkers after single oral doses of the anticoagulant agents dabigatran etexilate and rivaroxaban in healthy young male subjects and in healthy elderly subjects.

ELIGIBILITY:
Inclusion criteria for non-hemophilia participants:

Panel A

- Male or female between 65 to 85 years of age

Panel B

- Male between 18 to 45 years of age

Both Panels

* Weight of ≥50 kg and ≤110 kg
* In good health
* No clinically significant abnormality on electrocardiogram (ECG)
* Nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months

Exclusion criteria for non-hemophilia participants:

* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal (including peptic ulcer disease), cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* History of malignant neoplastic disease, with the exception of adequately treated non-melanomatous skin carcinoma or other malignancies that have been successfully treated ≥10 years prior to the study
* History of a thrombotic or platelet-related disorder including prior deep venous thrombosis or pulmonary embolus
* Use of warfarin, coumadin, heparin, aspirin, dabigatran etexilate, rivaroxaban or dipyridamole within 2 weeks
* History of poor wound healing
* Unable to refrain from or anticipates the use of any medication, including aspirin and aspirin-containing products, all non-steroidal anti-inflammatory drug (NSAID)-containing products (including pain, cold and allergy products, etc.) and including prescription and non-prescription drugs or herbal remedies (such as St. John's Wort [Hypericum perforatum]) beginning approximately 2 weeks (or 5 half-lives) prior to initiation of the treatment periods, throughout the study until the post-study visit
* Consumption of excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day
* Consumption of excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day
* Major surgery, donation or loss of 1 unit of blood (approximately 500 mL) or participation in another investigational study within 4 weeks
* History of significant multiple and/or severe allergies (including latex allergy), or an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food, including dabigatran etexilate and rivaroxaban
* Current regular user (including illicit drugs or has a history of drug [including alcohol] abuse within approximately 6 months
* History (including family history if hereditary) or symptoms of clinically relevant bleeding disorder
* Organic lesion at risk of bleeding (e.g., aneurysm, cavernous hemangioma, arterio-venous malformation)
* History of frequent epistaxis or has recurrent or active gingivitis or hemorrhoids

Inclusion criteria for hemophilia participants:

* Male with diagnosis of hemophilia B between 18 to 64 years of age
* Weight of ≥110 lbs and ≤300 lbs
* Has not received clotting factor in the 7 days prior to blood sampling
* No active bleeding event
* No procedure or surgery in the past 8 weeks
* Judged to be in good health based on medical history
* Has not smoked more than 2 cigarettes per day for at least approximately 1 week prior; has not smoked a pipe or cigar or chewed tobacco for at least 3 days prior
* Can refrain from the use of all NSAIDs (e.g., Advil, Aleve, aspirin), all NSAID-containing products (including pain, cold, and allergy products, etc.), herbal meds or drugs for 7 days prior to the date of study procedure

Exclusion criteria for hemophilia participants:

* Clinically significant endocrine, gastrointestinal (including peptic ulcer disease), cardiovascular, hematological (except factor IX deficiency), immunological, renal, respiratory, neurological or genitourinary abnormalities or diseases
* History of malignant neoplastic disease, with the exception of adequately treated non-melanomatous skin carcinoma or other malignancies that have been successfully treated ≥10 years prior to the study
* Consumption of excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) within 24 hours prior to study procedures
* Major surgery, donation or loss of 1 unit of blood (approximately 500 mL) or participation in another investigational study within 7 days prior to the date of study procedures
* Current regular user (including illicit drugs or has a history of drug [including alcohol] abuse within approximately 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Endogenous thrombin potential by Thrombin Generation Assay (TGA)-2a assay | From up to 2 hours pre-dose to up to 24 hours post-dose
Level of fibrin degradation product (D-dimer) | From up to 2 hours pre-dose to up to 24 hours post-dose
Level of fibrinopeptide A (FPA) | From up to 2 hours pre-dose to up to 24 hours post-dose
Level of prothrombin split products (F1+2) | From up to 2 hours pre-dose to up to 24 hours post-dose
Level of thrombin-antithrombin complex (TAT) | From up to 2 hours pre-dose to up to 24 hours post-dose